CLINICAL TRIAL: NCT06426251
Title: A Randomized Trial of Photobiomodulation Effect in Patients Receiving Total Knee Arthroplasty
Brief Title: Photobiomodulation Therapy in Patients Receiving Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111-036-F
Record Dates: First submitted 2022-08-02; First posted 2024-05-23 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Inflammation; Osteoarthritis; Post Operative Pain
MeSH Terms: conditions — Inflammation; Osteoarthritis; Pain, Postoperative | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): This group of patient will receive photobiomodulation pads on the part of surgical site and the machine will emit near-infrared light.
  Interventions: Device: Photobiomodulation
- control group (Sham Comparator): This group of patient will have photobiomodulation pads on the body surface as intervention group, but the machine will not emit near-infrared light.
  Interventions: Device: Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — Photobiomodulation therapy will be given daily start on the first day after surgery to post operative day 6

SUMMARY:
Photobiomdoulation is the use of near-infrared light to relieve pain, stimulate healing and reduce inflammation. Swelling and inflammation is a common condition after orthopedics surgeries over extremity and spine. This study aim to evaluate the effect of photobiomodulation over patients after Total Knee Arthroplasty.

DETAILED DESCRIPTION:
Patients aged over 20 after Total Knee Arthroplasty in our institution would be candidate for recruitment. The patients will be randomized to receive routine post operative care or photobiomodulation therapy. The swelling extent and subjective outcome will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* total knee arthroplasty

Exclusion Criteria:

* open injury
* pregnancy
* wound without primary closure
* infection
* previous surgery over surgical site
* skin defect

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
the change of bioimpedance | the bioimpedance measured once daily since post operative day1 to day6 and at 2 weeks
  bioimpedance of the surgical site will be measured for evaluation of swelling change

SECONDARY OUTCOMES:
pain score (visual analogue score) | once daily since post operative day1 to day6
  patient reported pain score, from 0 to 100 points
active range of motion of knee | once daily since post operative day1 to day6
  active range of motion of knee
2 minute walk test | once daily since post operative day1 to day6
  the distance that the patient could walk within 2 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Chieh Hsieh, Study Chair — National Taiwan University Hospital Hsin-Chu Branch
Locations (1):
- National Taiwan University Hospital, Hsin-Chu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Rezende MU, Varone BB, Martuscelli DF, Ocampos GP, Freire GMG, Pinto NC, de Sousa MVP. Pilot study of the effect of therapeutic photobiomodulation on postoperative pain in knee arthroplasty. Braz J Anesthesiol. 2022 Jan-Feb;72(1):159-161. doi: 10.1016/j.bjane.2021.07.040. Epub 2021 Nov 17. PMID 34800495
- [Background] Vassao PG, Renno AC, Smith BN, Bennett GB, Murphy M, Liebert A, Chow R, Laakso EL. Pre-Conditioning and Post-Operative Photobiomodulation Therapy by a Novel Light Patch System for Knee Arthroplasty: A Protocol for a Phase 1 Study. Photobiomodul Photomed Laser Surg. 2020 Apr;38(4):206-214. doi: 10.1089/photob.2019.4751. Epub 2020 Mar 18. PMID 32186975
- [Derived] Chia WT, Wong TH, Jaw FS, Hsieh HC. The Impact of Photobiomodulation Therapy on Swelling Reduction and Recovery Enhancement in Total Knee Arthroplasty: A Randomized Clinical Trial. Photobiomodul Photomed Laser Surg. 2025 Feb;43(2):65-72. doi: 10.1089/photob.2024.0120. Epub 2025 Jan 9. PMID 39786308